CLINICAL TRIAL: NCT01213888
Title: Trientine Hydrochloride for the Prevention of Macular Edema Associated With Pan-retinal Photocoagulation for Severe Non-proliferative and Proliferative Diabetic Retinopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment & superior treatments available for diabetic macular edema including anti-VEFG therapies such as bevacizumab and ranibizumab.
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: H08-01900
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic retinopathy; pan-retinal photocoagulation; macular edema
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Trientine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm II (Experimental)
  Interventions: Drug: Trientine Hydrochloride
- Arm I. Placebo + Pan-Retinal Photocoagulation (Placebo Comparator): All participating subjects will all receive PRP (pan-retinal photocoagulation) according to present standards of care; however, subjects randomized the placebo group will be on a 10-day course of oral placebo capsules at 1500mg administered for 7-days prior to and 3 days after the PRP sessions.
  Interventions: Drug: Oral placebo capsules

INTERVENTIONS:
Drug: Trientine Hydrochloride — All participating subjects will all receive PRP (pan-retinal photocoagulation) according to present standards of care; however, subjects randomized the intervention group (trientine hydrochloride) will be on a 10-day course of oral Trientine at 1500mg administered for 7-days prior to and 3 days after the PRP sessions.
  Other Names: Syprine
  Arms: Arm II
Drug: Oral placebo capsules — All participating subjects will all receive PRP (pan-retinal photocoagulation) according to present standards of care; however, subjects randomized the placebo group will be on a 10-day course of oral placebo capsules at 1500mg administered for 7-days prior to and 3 days after the PRP sessions
  Arms: Arm I. Placebo + Pan-Retinal Photocoagulation

SUMMARY:
To evaluate the effects of Trientine Hydrochloride in prevention of post-laser (pan-retinal photocoagulation) macular edema in the eyes for subjects with diabetic retinopathy. Trientine hydrochloride can limit secondary inflammatory damage to retinal vessels following the administration of pan-retinal photocoagulation therapy for severe non-proliferative diabetic retinopathy or retinal neovascularization due to diabetic retinopathy, resulting in less macular edema and improved visual outcomes.

DETAILED DESCRIPTION:
Individuals with new-onset severe non-proliferative diabetic retinopathy or retinal neovascularization who present to the retinal service of the UBC/VGH Eye Care Centre will be offered participation in this study. Subject inclusion criteria will parallel those of the DRS (Diabetic Retinopathy Study) and ETDRS (Early Treatment of Diabetic Retinopathy Study). One PRP session will consist of between 800 to 1000 laser burns. Subjects with discomfort during laser (a known side-effect) will be treated with local anesthetics.

As noted, participating subjects will all receive PRP according to present standards of care; however, subjects will be randomized to either a 10-day course of oral Trientine at 1500mg administered for 7-days prior to and 3 days after the PRP sessions, or a placebo. Serum copper levels and urinary copper levels will be evaluated before and after Trientine administration to determine the amount of free copper present systemically at the time of PRP treatment.

Ocular outcomes will include visual acuity testing (ETDRS), fluorescein angiography and ocular coherence tomography (OCT). These studies will be used to evaluate retinal morphology and photoreceptor function pre and post laser. All these evaluations are considered part of the routine evaluation of diabetic retinopathy in subjects being treated with PRP.

Outcome measures will be assessed at day 2-post laser, week 1, and Day 28-30. Further clinical PRP treatment will be administered if necessary after Day 28-30 at the discretion of the patients' ophthalmologist.

The primary analysis will involve comparing the retinal thickness measurements between subjects undergoing PRP with and without Trientine use. Secondary analyses will involve evaluations of visual acuity and fluorescein angiography. As well, changes in visual acuity, angiographic leakage, and retinal thickness will be regressed against serum copper levels. Sample size calculations suggest 15 subjects per arm should be adequate to demonstrate a 40% reduction in retinal thickness with a power of 80% comparing subjects receiving Trientine to controls.

Subjects who are randomized to Trientine will receive 1500 mg Trientine PO daily for 10 days. Subjects, study-coordinators, and investigators will be masked to treatment group. The primary analysis will be a comparison of OCT thickness measurements.

This is a single centre study involving 30 subjects (15 cases and 15 controls). A 1:1 randomization will be employed (Trientine 1500 mg: Placebo). No normal subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Severe non-proliferative diabetic retinopathy or retinal neovascularization secondary to diabetic retinopathy meeting DRS criteria for PRP laser
* ETDRS (Early treatment of Diabetic Retinopathy Study) eye score of at least 34-73 letters (at 2 meters) (20/20 to 20/320) for study eye and 20/800 in non-study eye
* Clinical evidence of macular microantiopathy in the study eye (lipid or retinal thickness is acceptable)
* No other ocular disease that could be responsible for decreased vision, macular edema or could limit macular imaging

Exclusion Criteria:

* Individuals with retinal neovascularization from causes other than diabetic retinopathy
* Any intraocular surgery within 2 months or Yag capsulotomy within 1 month in the study eye
* Prior retinal or vitreous surgery (including posterior segment vitrectomy or scleral buckling)
* Medical conditions requiring the use of mineral supplements (copper in particular)
* Individuals with anemia
* Individuals with mental or physical disabilities that prevent accurate vision testing
* History of treatment of PDR by PRP
* Active hepatitis, clinically significant liver disease or any evidence of renal failure.
* Stroke or myocardial infarction within preceding 6 months or ventricular tachycardia under treatment
* History of severe cardiac disease or unstable angina
* Subjects who are in an experimental therapy study or who have received experimental therapy within the last 12 weeks
* Subjects who are a poor medical risk because of other systemic diseases or active uncontrolled infections
* Women of childbearing potential not on 2 effective forms of birth control
* Women who are pregnant or plan to become pregnant
* Subjects with an allergy to fluorescein dye.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of a copper chelator in suppressing post-PRP macular edema in eyes with retinal neovascularization.
  The treatment effect will be measured by assessing changes in photoreceptor function (via visual acuity and contrast sensitivity) as well as retinal inflammation and thickening (via Fluorescein Angiography and Ocular Coherence Tomography).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ma, Study Director — University of British Columbia; Andrew Merkus, Study Director — University of British Columbia; David Albiani, Study Director — University of British Columbia; David Maberly, Principal Investigator — University of British Columbia
Locations (1):
- Eye Care Centre - Vancouver Coastal Health, Vancouver, British Columbia, Canada